CLINICAL TRIAL: NCT02374047
Title: A 2-Part, Phase 1, Single and Multiple Ascending Dose Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of CAT-2054 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catabasis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CAT-2054-101
Record Dates: First submitted 2015-02-02; First posted 2015-02-27 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (12):
- Cohort A1, Dose Level 1: CAT-2054 or placebo fasting (Experimental): Single dose
  Interventions: Drug: CAT-2054; Drug: Placebo
- Cohort A2, Dose Level 2: CAT-2054 or placebo fasting and fed (Experimental): Single dose
  Interventions: Drug: CAT-2054; Drug: Placebo
- Cohort A3, Dose Level 3: CAT-2054 or placebo fasting and fed (Experimental): Single dose
  Interventions: Drug: CAT-2054; Drug: Placebo
- Cohort A4, Dose Level 4: CAT-2054 or placebo fasting and fed (Experimental): Single dose
  Interventions: Drug: CAT-2054; Drug: Placebo
- Cohort A5, Dose Level 5: CAT-2054-C or placebo fasting and fed (Experimental): Single dose
  Interventions: Drug: Placebo; Drug: CAT-2054-C
- Cohort B1, Dose Level 1: CAT-2054 or placebo (Experimental): Multiple dose for 14 days
  Interventions: Drug: CAT-2054; Drug: Placebo
- Cohort B2, Dose Level 2: CAT-2054 or placebo (Experimental): Multiple dose for 14 days
  Interventions: Drug: CAT-2054; Drug: Placebo
- Cohort B3, Dose Level 3: CAT-2054 or placebo (Experimental): Multiple dose for 14 days
  Interventions: Drug: CAT-2054; Drug: Placebo
- Cohort B4, Dose Level 4: CAT-2054 or placebo (Experimental): Multiple dose for 14 days
  Interventions: Drug: CAT-2054; Drug: Placebo
- Cohort B5, Dose Level 5: CAT-2054 or placebo (Experimental): Multiple dose for 14 days
  Interventions: Drug: CAT-2054; Drug: Placebo
- Cohort B6, Dose Level 6: CAT-2054 with atorvastatin (Experimental): Multiple dose for 14 days
  Interventions: Drug: CAT-2054; Drug: Atorvastatin
- Cohort B7, Dose Level 7: CAT-2054 or placebo (Experimental): Multiple dose for 14 days
  Interventions: Drug: CAT-2054; Drug: Placebo

INTERVENTIONS:
Drug: CAT-2054
  Arms: Cohort A1, Dose Level 1: CAT-2054 or placebo fasting; Cohort A2, Dose Level 2: CAT-2054 or placebo fasting and fed; Cohort A3, Dose Level 3: CAT-2054 or placebo fasting and fed; Cohort A4, Dose Level 4: CAT-2054 or placebo fasting and fed; Cohort B1, Dose Level 1: CAT-2054 or placebo; Cohort B2, Dose Level 2: CAT-2054 or placebo; Cohort B3, Dose Level 3: CAT-2054 or placebo; Cohort B4, Dose Level 4: CAT-2054 or placebo; Cohort B5, Dose Level 5: CAT-2054 or placebo; Cohort B6, Dose Level 6: CAT-2054 with atorvastatin; Cohort B7, Dose Level 7: CAT-2054 or placebo
Drug: Placebo
  Arms: Cohort A1, Dose Level 1: CAT-2054 or placebo fasting; Cohort A2, Dose Level 2: CAT-2054 or placebo fasting and fed; Cohort A3, Dose Level 3: CAT-2054 or placebo fasting and fed; Cohort A4, Dose Level 4: CAT-2054 or placebo fasting and fed; Cohort A5, Dose Level 5: CAT-2054-C or placebo fasting and fed; Cohort B1, Dose Level 1: CAT-2054 or placebo; Cohort B2, Dose Level 2: CAT-2054 or placebo; Cohort B3, Dose Level 3: CAT-2054 or placebo; Cohort B4, Dose Level 4: CAT-2054 or placebo; Cohort B5, Dose Level 5: CAT-2054 or placebo; Cohort B7, Dose Level 7: CAT-2054 or placebo
Drug: CAT-2054-C
  Arms: Cohort A5, Dose Level 5: CAT-2054-C or placebo fasting and fed
Drug: Atorvastatin
  Arms: Cohort B6, Dose Level 6: CAT-2054 with atorvastatin

SUMMARY:
This is a 2-part, Phase 1, placebo-controlled, double-blind, randomized, single and multiple ascending dose study. CAT-2054 will be administered either as an uncoated capsule (CAT-2054) or a coated capsule (CAT-2054-C). In Part A, CAT-2054 or placebo is administered as a single dose in a fasting state at 4 dose levels; at 3 dose levels, subjects will return for a second dose of the study drug after a high-fat meal. Additionally, at 1 dose level, CAT-2054-C or placebo will be administered as a single dose in a fasting state, and subjects will return for a second dose of the study drug after a high-fat meal. In Part B, CAT-2054 will be administered as multiple ascending doses at 4 dose levels for 14 consecutive days. In selected cohorts, CAT-2054, CAT-2054-C or CAT-2054 with atorvastatin will be dosed to assess safety in anticipation of future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent before any study-specific procedure
* Good health as determined by medical history, physical examination, vital sign measurements, ECG, and clinical laboratory measurements
* Satisfies one of the following:

  1. Females not of childbearing potential: non-pregnant and non-lactating surgically sterile or postmenopausal 2 years or less with a follicle-stimulating hormone assessment greater than or equal to 40 IU/L
  2. Males: surgically sterile, abstinent, or subject or partner is utilizing an acceptable contraceptive method during and 3 months after the last study dose
* For Part B only, measured at Screening: Fasting LDL-C ≥100 mg/dL; or (Cohort B6 only) fasting LDL-C ≥130 mg/dL
* Body mass index (BMI) between 18 and 30 kg/m², inclusive, for Part A and between 18 and 40 kg/m², inclusive, for Part B, and body weight >50 kg at Screening

Exclusion Criteria:

* Use of prescription drugs or non-prescription drugs including herbals, and dietary supplements (including multivitamins and any product containing niacin or omega-3 fatty acids above the Recommended Daily Allowance) within 2 weeks before dosing. Additionally for Part B only, use of any lipid-regulating prescription drug, non-prescription drug, herbal, or dietary supplement within 6 weeks before dosing
* Clinically significant disease that requires a physician's care and/or would interfere with study evaluations
* Clinically significant electrocardiogram (ECG) abnormalities or laboratory results as assessed by the investigator, such as QTcF >450
* Use of any investigational drug or participation in any investigational study within 30 days prior to screening or 5 half-lives of the study agent, whichever is longer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of adverse events | up to 3 weeks

SECONDARY OUTCOMES:
AUCinf of CAT-2054 | Days 1 through 4
Cmax of CAT-2054 | up to 3 weeks
Changes from baseline for hematology, chemistry, coagulation and urinalysis | up to 3 weeks
Assess the pharmacodynamic effects of multiple doses of CAT-2054 on serum lipids LDL-C, non-HDL-C, total cholesterol, triglycerides, HDL-C, apoB, and PCSK9. | up to 3 weeks
AUC48 of Atorvastatin | up to 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States